CLINICAL TRIAL: NCT02017041
Title: Using mHealth to Aid Opioid Medication Adherence Pilot Study
Status: Completed | Type: Observational
Sponsor: Care Team Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: HHSN271201300015C-1; HHSN271201300015C (Other Grant/Funding Number: National Institute on Drug Abuse (NIDA/NIH))
Record Dates: First submitted 2013-12-09; First posted 2013-12-20 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Opioid Dependence
Keywords: opioid dependence, buprenorphine, smartphone, suboxone
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- buprenorphine/naloxone: Opioid substitution therapy patient taking buprenorphine/naloxone, MedSignals and smartphone app.
  Interventions: Device: Medsignals; Device: smartphone app

INTERVENTIONS:
Device: Medsignals — MedSignals (www.medsignals.com) is a cellular communicating medication management device designed to improve adherence. It will be used to track when medication is removed from the device at dosing times and deliver audible and visual alerts at dosing times and to relay adherence data securely to patient files. Participants will use this device throughout the 5-week trial. It is a Class I device.
Device: smartphone app — The smartphone app being evaluated in this study is designed to support effective medication management of opioid substitution patients taking buprenorphine/naloxone.

SUMMARY:
The purpose of this study is to evaluate the usability of an interactive smartphone application (app) designed to engage and support patients receiving bup/nal.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the usability of a medication management aid for opioid dependence named SubAID. The SubAID system is a smartphone application and medication monitor designed to optimize adherence behaviors of an OD patient responsible for administering bup/nal maintenance therapy medication.

Usability of the SubAID system will be tested utilizing a 3-Stage study design over a 5 week period among a cohort of subjects prescribed bup/nal and undergoing OST.

* Stage 1 - 1 week: Participants will use only an electronic medication monitor (MedSignals) in control mode to passively record baseline adherence to medication.
* Stage 2 - 2 weeks: Participants will use MedSignals in control mode and the smartphone application.
* Stage 3 - 2 weeks: Participants will use MedSignals in active mode and the smartphone application.

After each stage usability assessments will be conducted to evaluate satisfaction with the products from participants.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age
* Physician diagnosis of opioid dependence (OD)
* Prescribed buprenorphine/naloxone (bup/nal) and acclimated to medication.
* Able to speak and read English
* Willing to provide written informed consent prior to study entry
* Able to understand the study
* Ownership of an Android or iPhone smartphone

Exclusion Criteria:

* Having any concurrent medical or psychiatric condition that, in the investigator's opinion, may preclude participation in this study; or
* Cognitive or other impairment that would interfere with completing a self-administered questionnaire.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
questionnaire assessing usability of the system. | up to 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bailey, PhD, Study Director — Care Team Solutions
Locations (1):
- Care Team Solutions, Lexington, Kentucky, United States